CLINICAL TRIAL: NCT03164434
Title: Influence of Drainage of Cerebrospinal Fluid on ICP Signals Obtained Through an External Ventricular Drain.
Brief Title: Influence of Drainage on EVD ICP-signal
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Bart Depreitere, professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: EVD-ICP
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Head Injury; Subarachnoid Hemorrhage
Keywords: intracranial pressure; cerebrospinal fluid drainage; waveform analysis
MeSH Terms: conditions — Craniocerebral Trauma; Subarachnoid Hemorrhage; Cerebrospinal Fluid Leak

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study investigates ICP signals obtained through an external ventricular drain in the brain connected with an external transducer. In particular, the study investigates how drainage influences the monitored signal: influence of flow rate, reservoir height and initial ICP before draining.

ELIGIBILITY:
Inclusion Criteria:

* TBI/SAH patients with need for ICP monitoring

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe traumatic brain injury or subarachnoid hemorrhage in whom monitoring of ICP is warranted.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
ICP signal changes | immediate during drainage
  changes in magnitude and amplitude of ICP pulse during drainage of CSF

CONTACTS AND LOCATIONS:
Overall Officials: Bart Depreitere, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium